CLINICAL TRIAL: NCT02663271
Title: A Phase 2, Multi-center, Single Arm, Histologically Controlled Study Testing the Combination of TTFields and Pulsed Bevacizumab Treatment in Patients With Bevacizumab-refractory Recurrent Glioblastoma
Brief Title: TTFields and Pulsed Bevacizumab for Recurrent Glioblastoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: stagnant enrollment
Sponsor: University of Florida (Other)
Collaborators: NovoCure Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB201600074; OCR14874 (Other: University of Florida)
Record Dates: First submitted 2016-01-21; First posted 2016-01-26 (Estimated); Results first posted 2022-06-23 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-05

CONDITIONS: Glioblastoma Multiforme; Glioblastoma; Malignant Glioma; GBM
MeSH Terms: conditions — Glioblastoma; Glioma | interventions — Bevacizumab; Magnetic Resonance Spectroscopy; Karnofsky Performance Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Optune+Pulsed Bevacizumab (Experimental): The subjects will undergo 12 months of planned continuous treatment with Optune. The treatment will begin at week 0 and will be continuous throughout the study. Pulsed bevacizumab dosing is defined by at least one cycle on and at least one cycle off. A cycle is defined as 8 weeks in length. If after one cycle on, there is no evidence of a repeat response; bevacizumab will be continued for one more cycle. If after two cycles on, there is no repeat response; bevacizumab will be continued with or without other standard chemotherapy until death. If after at least one cycle on, there is evidence of repeat response, bevacizumab will be discontinued for at least one cycle. In addition, the following will be performed: Bevacizumab will be given, physical examination and quality of life questionnaires will be performed and brain MRI.
  Interventions: Drug: Bevacizumab; Device: Optune; Other: Brain MRI; Other: Quality of Life Questionnaires

INTERVENTIONS:
Drug: Bevacizumab — Bevacizumab will be given at 10mg/kg IV every 2 weeks.
  Other Names: Avastin
Device: Optune — Optune will be worn continuously for 12 months. Optune is programmed by Novocure to deliver 200 kHz TTFields in two sequential, perpendicular field directions at a maximal intensity of 707mARMS. There will be no adjustments made to the device by investigators or patients/caregivers.
  Other Names: NovoTTF™-100A System
Other: Brain MRI — Brain MRI will be done at screening and every 8 weeks.
  Other Names: Magnetic resonance imaging
Other: Quality of Life Questionnaires — The quality of life questionnaires will be performed within 14 days of treatment and every 4 weeks.
  Other Names: Karnofsky Performance Scale; MMSE

SUMMARY:
Glioblastoma multiforme (GBM) is the most common and deadliest primary malignant neoplasm of the central nervous system in adults. Despite an aggressive multimodality treatment approach including surgery, radiation therapy and chemotherapy, overall survival remains poor. Novocure has shown that when properly tuned, very low intensity, intermediate frequency electric fields (TTFields) stunt the growth of tumor cells. The Optune system (NovoTTFTM Therapy) is a portable battery operated device, which produces TTFields within the human body by means of surface transducer arrays. The TTFields are applied to the patient by means of surface transducer arrays that are electrically insulated, so that resistively coupled electric currents are not delivered to the patient. Optune is currently FDA-approved as a single modality treatment for recurrent GBM when both surgical and radiotherapy options have been exhausted as well as combination with adjuvant temozolomide for newly diagnosed GBM.

This research study is being performed to determine whether or not TTFields combined with pulsed bevacizumab treatment increases overall survival in patients with bevacizumab-refractory GBM compared to historical controls treated with continuous bevacizumab alone or in combination with other chemotherapy.

DETAILED DESCRIPTION:
Subjects who have evidence of bevacizumab-refractory GBM will be eligible to participate in this research study. Subjects will undergo 12 months of planned continuous treatment with TTFields followed by pulsed bevacizumab treatment when there is evidence of further progression per RANO, with the option of extending treatment up to a total of 24 months in patients who have not progressed and/or have adequate performance status at the 12 month mark. Pulsed bevacizumab dosing is defined by at least one cycle on and at least one cycle off. A cycle is defined as 8 weeks in length. If after one cycle on, there is no evidence of a repeat response; bevacizumab will be continued for one more cycle. If after two cycles on, there is no repeat response; bevacizumab will be continued with or without other standard chemotherapy until death. If after at least one cycle on, there is evidence of repeat response, bevacizumab will be discontinued for at least one cycle or until progression is noted again per RANO, whichever is later, at which time pulsed bevacizumab will be restarted as outlined above. The investigators believe that this approach will produce peaks and troughs in mitotic activities of glioma cells that render glioma cells more sensitive to the antimitotic activity of Optune during peak growth rates, thus lowering disease burden and increasing survival. In addition, the following will be performed: Bevacizumab will be given at 10mg/kg IV every 2 weeks. Physical examination and quality of life (QoL) assessments will be performed bi-monthly. Brain MRI will be performed every 2 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed GBM, WHO grade IV. GBM variants and secondary GBM are allowed in any recurrence (including multiple) and have been treated with radiation and chemotherapy.
* Unequivocal evidence of tumor progression during prior bevacizumab treatment per RANO criteria.
* Patient is a candidate for, and agrees to proceed with additional bevacizumab treatment.
* Male or female at least 22 years of age or older.
* Karnofsky Performance Scale (KPS) ≥ 60%.
* Planned treatment with TTFields therapy.
* Women of childbearing potential must have a negative serum or urine pregnancy test within 14 days of treatment.
* Participants of childbearing/reproductive potential must use effective contraception.
* Participants must be able to understand and willing to comply with protocol requirements as assessed by the investigator.
* Signed informed consent according to institutional guidelines prior to registration.

Exclusion Criteria:

* Inability to undergo brain MRI due to medical or personal reasons.
* Currently receiving investigational agents that are intended as treatments of recurrent GBM.
* Skull defect such as missing bone or bullet fragments.
* Uncontrolled intercurrent illness including, but not limited to symptomatic congestive heart failure, unstable angina pectoris, heart attack within the previous 12 months, stroke (except for TIA) within the previous 6 months, or psychiatric illness/social situations that would limit compliance with study requirements.
* Intracranial hemorrhage except for tumor associated micro hemorrhage.
* Women who are pregnant or breastfeeding.
* Implanted pacemaker, programmable shunts, defibrillator, deep brain stimulator, vagus nerve stimulator, and other implanted electronic devices in the brain or the spinal cord.
* Tumor located entirely in the infratentorium.
* History of hypersensitivity to hydrogel.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-12-19 (Actual); Primary Completion 2021-06-11 (Actual); Study Completion 2021-06-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David D Tran, MD, PhD, Principal Investigator — University of Florida
Locations (2):
- United States (2):
  - University of Florida, Gainesville, Florida
  - Washington University, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Ten patients were assessed for eligibility in this study. One subject did not meet eligibility.
Period: Overall Study
Arm/Group | Optune+Pulsed Bevacizumab
Started | 9
Completed | 3
Not Completed | 6
Not completed — Withdrawal by Subject | 5
Not completed — Lack of Efficacy | 1

BASELINE CHARACTERISTICS:
Arm/Group | Optune+Pulsed Bevacizumab
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.7 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Overall survival is defined as time interval from date of starting Optune to date of death or censoring whichever happens first.
Time Frame: from date of starting Optune to date of death or censoring, whichever comes first, assessed up to 24 months
Population: participants completing at least 8 weeks of treatment with the Optune device with compliance rate > 60% in at least one 4-week period
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Optune+Pulsed Bevacizumab
Number analyzed (Participants) | 3
months | 7.4 [5 to NA] — insufficient number of participants with events
Statistical Analysis 1: Comparison: Optune+Pulsed Bevacizumab; Test type: Superiority — We used one-sample log rank test to compare to historical control; p < 0.001, Log Rank; Hazard Ratio (HR) = 0.3

2. Secondary Outcome: Karnofsky Performance Scale
Description: The Karnofsky Performance Scale is rated from 0 - 100 with 0 = death and 100 = normal without complaints or evidence of disease. A higher score means the patient is better able to carry out daily activities. Patients are evaluable for assessment of QoL after completing at least 8 weeks of treatment with the Optune device with compliance rate > 60% in at least one 4-week period.
Time Frame: Assessed up to 24 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Optune+Pulsed Bevacizumab
Number analyzed (Participants) | 3
score on a scale | 73.3 (5.8)

3. Secondary Outcome: Mini-Mental Status Exam
Description: The Mini Mental State Examination (MMSE) it is an 11-question measure that tests five areas of cognitive function: orientation, registration, attention and calculation, recall, and language. The maximum score is 30. The higher the score suggests less cognitive impairment. A score of 24-30 suggests no cognitive impairment. A score of 18-23 suggests mild cognitive impairment. A score of 0-17 suggests severe cognitive impairment. Patients are evaluable for assessment of QoL after completing at least 8 weeks of treatment with the Optune device with compliance rate > 60% in at least one 4-week period.
Time Frame: Assessed up to 24 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Optune+Pulsed Bevacizumab
Number analyzed (Participants) | 3
score on a scale | 23.2 (5.1)

4. Secondary Outcome: Response Assessment in Neuro-Oncology (RANO) Measurement Form
Description: The Response Assessment in Neuro-Oncology criteria were developed as an objective tool for radiologic assessment of treatment response in high-grade gliomas. Disease progression is defined as ≥ 25% increase in sum of the products of perpendicular diameters of enhancing lesions (with the absolute increase of at least 1 dimension of at least 5 mm) compared with the smallest tumor measurement obtained either at baseline. Response assessment will be performed for patients completing at least 8 weeks of treatment with the Optune device with compliance rate > 60% in at least one 4-week period.
Time Frame: Assessed up to 24 months
Population: after completing at least 8 weeks of treatment with the Optune device with compliance rate > 60% in at least one 4-week period.
Measure: Count of Participants; unit: Participants
Arm/Group | Optune+Pulsed Bevacizumab
Number analyzed (Participants) | 3
Participants
  Progressive disease | 2
  Stable disease | 1

ADVERSE EVENTS:
Time Frame: Adverse events were collected from start of treatment with Optune and continuously throughout study treatment (up to 24 months) plus an additional 30 days post study completion or withdrawal for up to 25 months.
Arm/Group | Optune+Pulsed Bevacizumab
All-Cause Mortality (participants affected / at risk) | 6/9
Serious Adverse Events (participants affected / at risk) | 4/9
Other Adverse Events (participants affected / at risk) | 6/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Optune+Pulsed Bevacizumab (N=9)
Non-cardiac chest pain (General disorders) | 1 (1)
thromboembolic event (Vascular disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Nervous system disorder (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Optune+Pulsed Bevacizumab (N=9)
Confusion (Psychiatric disorders) | 4 (6)
Anxiety (Psychiatric disorders) | 2 (6)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (4)
Seizure (Nervous system disorders) | 5 (8)
Depression (Psychiatric disorders) | 2 (4)
Fatigue (General disorders) | 3 (3)
Memory impairment (Nervous system disorders) | 1 (1)
Blurred vision (Eye disorders) | 1 (2)
Dysphasia (Nervous system disorders) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 2 (3)
Extremity pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (2)
Dizziness (Nervous system disorders) | 1 (1)
Dysarthria (Nervous system disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Edema (General disorders) | 2 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 1 (1)
Intracranial hemorrhage (Nervous system disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (2)
Vomiting (Gastrointestinal disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Platelet count decreased (Investigations) | 1 (2)
Nervous System Disorder (Nervous system disorders) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-15): https://cdn.clinicaltrials.gov/large-docs/71/NCT02663271/Prot_SAP_000.pdf